CLINICAL TRIAL: NCT01260051
Title: Intrapartum Epidural Fentanyl/Bupivacaine Analgesia, Infant Feeding Behavior, & Breast-Feeding Outcomes
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: uhcmc
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia, Epidural; Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidural Recipients
- Non-Epidural Recipients

SUMMARY:
Currently, no clear consensus exists regarding the effect of epidural anesthesia upon breast-feeding. In theory, epidurals may increase breast-feeding failure via inadequate maternal milk production, deficiencies in neonatal neurobehavior, or both, but most studies have failed to separate these potential mechanisms. The present study examines whether epidural duration correlates with 1) likelihood of breast-feeding at hospital discharge and 2) neonatal neurobehavioral deficits in feeding, as measured by the L&A components of the standardized, validated LATCH scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery
* Delivery of a single live neonate

Exclusion Criteria:

* NICU admission following delivery
* Pitocin augmentation

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Parturients who delivered at UHCMC between August 2009 and January 2010
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Breast-Feeding at Hospital Discharge | Baseline
  This outcome variable is binary. If a woman is breast-feeding with bottle supplementation at the time of hospital discharge, then she is recorded as "Yes."

SECONDARY OUTCOMES:
L&A Components of LATCH Score | Baseline
  The L component of the score measures neonatal ability to latch at the breast and the A component measures the presence of audible swallows, which are variables that reflect neonatal neurobehavioral capacity with respect to feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L Szabo, MD Candidate, Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Kumar SP, Mooney R, Wieser LJ, Havstad S. The LATCH scoring system and prediction of breastfeeding duration. J Hum Lact. 2006 Nov;22(4):391-7. doi: 10.1177/0890334406293161. PMID 17062784
- [Background] Beilin Y, Bodian CA, Weiser J, Hossain S, Arnold I, Feierman DE, Martin G, Holzman I. Effect of labor epidural analgesia with and without fentanyl on infant breast-feeding: a prospective, randomized, double-blind study. Anesthesiology. 2005 Dec;103(6):1211-7. doi: 10.1097/00000542-200512000-00016. PMID 16306734
- [Background] Wiklund I, Norman M, Uvnas-Moberg K, Ransjo-Arvidson AB, Andolf E. Epidural analgesia: breast-feeding success and related factors. Midwifery. 2009 Apr;25(2):e31-8. doi: 10.1016/j.midw.2007.07.005. Epub 2007 Nov 5. PMID 17980469